CLINICAL TRIAL: NCT06194448
Title: A Phase II, Open-label, Single-arm Study of Osimertinib as Induction Therapy Prior to CRT and Maintenance Osimertinib in Patients With Epidermal Growth Factor Receptor (EGFR) Mutation-positive, Stage III, Unresectable Non-small Cell Lung Cancer (NEOLA)
Brief Title: To Evaluate the Efficacy/Safety of Osimertinib Prior to CRT and Maintenance of it With Stage III, Unresectable NSCLC With EGFR Mutations
Acronym: NEOLA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D516AC00003; 2023-507798-16-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-12-20; First posted 2024-01-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer
Keywords: EGFR +; Unresectable Non-small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — osimertinib; Cisplatin; Carboplatin; Pemetrexed; Paclitaxel; Radiation

STUDY DESIGN:
Intervention Model Description: Patients will receive open-label osimertinib induction treatment for 8 weeks (± 1 week window to account for patient variability and CRT scheduling), followed by CRT treatment for 6 weeks (± 1 week) and then osimertinib maintenance treatment until RECIST 1.1-defined radiological progression by investigator unless there is evidence of unacceptable toxicity or if the patient requests to stop the study treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label Osimertinib Induction Treatment (Experimental): Patients will receive open-label osimertinib induction treatment for 8 weeks (± 1 week window to account for patient variability and CRT scheduling), followed by CRT treatment for 6 weeks (± 1 week) and then osimertinib maintenance treatment until RECIST 1.1-defined radiological progression by investigator unless there is evidence of unacceptable toxicity or if the patient requests to stop the study treatment.
  Interventions: Drug: Osimertinib; Drug: Cisplatin or Carboplatin; Pemetrexed or Paclitaxel; Drug: Radiation

INTERVENTIONS:
Drug: Osimertinib — 80 mg daily (or 40 mg daily for dose reduction)
  Other Names: Tagrisso, AZD9291
Drug: Cisplatin or Carboplatin; Pemetrexed or Paclitaxel — Pemetrexed (500 mg/m2 to be administered on Day 1 of every 3-week cycle for 2 cycles) or Paclitaxel (175 mg/m2 on Day 1 of every 3-week cycle for 2 cycles) PLUS Cisplatin (75 mg/m2) or Carboplatin (AUC5) to be administered on Day 1 of every 3--week cycle for 2 cycles
Drug: Radiation — Patients must have received a total dose of radiation of 60 Gy ± 10% (54 to 66 Gy) as part of the chemoradiation therapy. It is recommended but not required that patients have a:
  * Mean lung dose < 20 Gy and/or V20 < 35%
  * Mean oesophagus dose < 34 Gy
  * Heart V50 < 25%, V30 < 50%, and V45 < 35%

SUMMARY:
The purpose of this study is to measure efficacy and safety of osimertinib as induction therapy prior to curative intent CRT and maintenance osimertinib in adult patients with Stage III, unresectable NSCLC with common EGFR mutations (exon 19 deletion or L858R).

DETAILED DESCRIPTION:
The study duration will be approximately 2 years for recruitment and 2 years of follow-up from the last patient's initiation into the study.

The induction treatment with osimertinib will be up to 8 weeks, followed by 6 weeks of CRT treatment and osimertinib maintenance treatment until PD or death.

The visit frequency will be every 2 weeks to 4 weeks during the induction treatment period, every 3 weeks during the CRT period (every 3 weeks for chemotherapy and daily visits for RT), and every 12 weeks during the osimertinib maintenance treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 or the legal age of consent in the jurisdiction in which the study is taking place, at the time of signing the informed consent form.
2. Patients with histologically documented NSCLC of predominantly non-squamous, squamous, and adenosquamous pathology who present with locally advanced, unresectable (Stage III) disease (according to Version 8 of the IASLC Staging Manual in Thoracic Oncology). It is recommended but not required that except for overt cT4 disease, nodal status N2, or N3 should have been proven by biopsy, via endobronchial ultrasound, mediastinoscopy, thoracoscopy, or in absence of biopsy, should have been confirmed with whole body 18FDG PET plus contrast-enhanced CT in addition to or in combination with PET.
3. Patient who are eligible for and - planning to undergo CCRT or SCRT treatment.
4. Patients who had recurred from Stage I/II/III after complete surgery or had gross incomplete resections can be included if they didn't receive treatment with any chemotherapy, radiation therapy, immunotherapy, targeted therapy, or investigational agents.
5. Patients with HBV are only eligible for inclusion if they meet all the following criteria:

   * Demonstrate absence of HCV co-infection or history of HCV co-infection
   * Demonstrate absence of HIV co-infection
   * Patients with active HBV infection are eligible if they are:

     * Receiving anti-viral treatment for at least 6 weeks prior to study treatment, HBV DNA is suppressed to <100 IU/mL and transaminase levels are below ULN.

   Participants with a resolved or chronic HBV infection are eligible if they are:
   * Negative for HBsAg and positive for hepatitis B core antibody [anti-HBc IgG or total anti-HBc Ab]. In addition, patients must be receiving anti-viral prophylaxis for 2-4 weeks prior to study treatment or
   * Positive for HBsAg, but for > 6 months have had transaminases levels below ULN and HBV DNA levels below <100 IU/mL (i.e., are in an inactive carrier state). In addition, patients must be receiving anti-viral prophylaxis for 2-4 weeks prior to study treatment.
6. Patients with HIV are only eligible for inclusion if they meet all the following criteria:

   * Demonstrate absence of HBV/ HCV co-infection
   * Undetectable viral RNA load for 6 months
   * CD4+ count of >350 cells/μL
   * No history of AIDS-defining opportunistic infection within the past 12 months
   * Stable for at least 4 weeks on the same anti-HIV medications
7. Availability of the EGFRm test results confirming that the tumour harbours one of the two common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R), either alone or in combination with other EGFR mutations including de novo T790M
8. WHO performance status of 0 or 1 with no deterioration over the previous 2 weeks prior to baseline at screening and prior to first dose.
9. Minimum life expectancy of > 12 weeks at Day 1.
10. At least one lesion that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes, which must have short axis ≥ 15 mm) with CT or MRI and is suitable for accurate repeated measurements.
11. Male and/or female. Contraceptive use by males or females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies and/or SoC CRT
12. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this CSP.
13. Provision of signed and dated written Optional Genomics Initiative Research Information and Consent Form prior to collection of samples for optional genomics initiative research that supports the Genomic Initiative.

Note: If a patient declines to participate in optional genetic research, there will be no penalty or loss of benefit to the patient, and he/she will not be excluded from other aspects of the study.

Exclusion Criteria:

1. Any presence of small cell and mixed small-cell and non-small cell histology.
2. Past medical history of ILD/pneumonitis, drug-induced ILD, radiation pneumonitis that required steroid treatment, or any evidence of clinically active ILD/pneumonitis.
3. Any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study treatment with the exception of alopecia and Grade 2 prior platinum-therapy related neuropathy. Patients with irreversible toxicity that is not reasonably expected to be exacerbated by study intervention in the opinion of the investigator may be included after consultation with the AstraZeneca medical monitor (eg, hearing loss).
4. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or active infection (eg, patients receiving treatment for infection, including HCV, HIV, and tuberculosis) or active uncontrolled HBV infection.
5. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib.
6. History of another primary malignancy except for malignancy treated with curative intent with no known active disease ≥ 2 years before the first dose of study intervention and of low potential risk for recurrence. Exceptions include adequately resected non-melanoma skin cancer and curatively treated in situ disease. Patients who have received RT with overlapping fields (eg, cured breast cancer) should be excluded.
7. Patient meets any of the following cardiac criteria:

   1. Mean resting QTc > 470 msec, obtained from 3 ECGs, using the screening clinic ECG machine-derived QTc value.
   2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG eg, complete left bundle branch block, third degree heart block and second-degree heart block. Patients with atrial fibrillation controlled by medication or arrhythmias controlled by pacemakers may be permitted based on the investigator judgement with cardiologist consultation recommended.
   3. History of QT prolongation associated with other medications that required discontinuation of that medication.
8. Congenital long QT syndrome, family history of long QT syndrome, unexplained sudden death under 40 years of age in first-degree relatives or patients with any factors that increase the risk of QTc prolongation/arrhythmic events such as electrolyte abnormalities, heart failure or any concomitant medication known to prolong the QT interval and cause TdP.
9. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

   * Absolute neutrophil count <1.5 × 10^9/L
   * Platelet count <100 × 10^9/L
   * Haemoglobin <90 g/L
   * Alanine transferase >2.5 times the upper limit of normal (ULN)
   * Aspartate transferase >2.5 times ULN
   * Total bilirubin >1.5 times ULN or >3 times ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia)
   * Creatinine >1.5 times ULN concurrent with creatinine clearance <50 mL/min (measured or calculated by Cockcroft and Gault formula); confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.
10. Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of CYP3A4 (at least 3-week prior to dosing). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4.
11. Prior treatment with any chemotherapy, radiation therapy, immunotherapy or investigational agents for locally advanced, unresectable Stage III NSCLC. Prior surgical resection (ie, Stage I, II, or III) with no systemic treatment with residual disease or a recurrence is permitted.
12. Prior exposure to EGFR-TKI therapy
13. Major surgical procedure (excluding placement of vascular access) or significant traumatic injury within 4 weeks of the first dose of study intervention or an anticipated need for major surgery during the study.
14. Participation in another clinical study with a study intervention or investigational medicinal device administered in the last 4 weeks (unless the safety profile is known prior to first dose of study intervention), or concurrent enrolment in another clinical study (unless the study is observational [noninterventional], or the patient is in the followup period of an interventional study).
15. History of hypersensitivity to active or inactive excipients of osimertinib or drugs with a similar chemical structure or class to osimertinib.
16. History of hypersensitivity to active or inactive excipients of the chemotherapy regimen of choice (pemetrexed or paclitaxel; cisplatin or carboplatin) or RT or drugs with a similar chemical structure or class to the chemotherapy.
17. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
18. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
19. Previous enrolment in the present study. Rescreening of individuals who were screen failures is allowed.
20. For females only: Currently pregnant (confirmed with positive pregnancy test) or breastfeeding.
21. Patients should refrain from breastfeeding from enrolment throughout the study and until 6 weeks after last dose of study intervention.
22. In addition, the following are considered criteria for exclusion from the exploratory genetic research:

    * Prior allogeneic bone marrow transplant.
    * Non-leukocyte depleted whole blood transfusion within 120 days of genetic sample collection.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2024-04-21 (Actual); Primary Completion 2026-07-07 (Estimated); Study Completion 2027-07-07 (Estimated)

PRIMARY OUTCOMES:
PFS (Progression-Free Survival) | Assessed from date of first dose to progression (up to a maximum of approximately 4 years)
  PFS is defined as the time from date of first dose until progression per RECIST 1.1 as assessed by the investigator at the local site, or death due to any cause.

SECONDARY OUTCOMES:
ORR (Objective Response Rate) | Assessed during the induction phase of the study, scans are carried out at baseline and week 8 (plus or minus visit window).
  ORR is defined as the proportion of patients who have a CR or PR, as determined by the investigator at local site per RECIST 1.1.
DCR (Disease Control Rate) | Assessed during the induction phase of the study, scans are carried out at baseline and week 8 (plus or minus visit window).
  DCR is defined as the percentage of subjects who have a best overall response of CR or PR or SD (at 8 weeks) as determined by the investigator at the local site per RECIST 1.1.
OS (Overall Survival) | Assessed from first dose to end of study or death (up to a maximum of approximately 4 years)
  OS is defined as time from date of first dose until the date of death due to any cause.
EFS (Event-Free Survival) | Assessed from first dose until a progression event or death (up to a maximum of approximately 4 years)
  EFS is defined as time from date of first dose until any of the following events: progression of disease that precludes CRT or completion of CRT, progression during or after CRT, or death due to any cause.

OTHER OUTCOMES:
AEs | from signing ICF to 28 days after last dose or end of study (up to a maximum of approximately 4 years)
  To assess the safety of osimertinib used as an induction therapy prior to CRT and maintenance osimertinib treatment by assessment of AEs in patients with unresectable EGFRm NSCLC

CONTACTS AND LOCATIONS:
Locations (35):
- United States (2):
  - Research Site, La Jolla, California
  - Research Site, Palo Alto, California
- China (12):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Zhengzhou
- Israel (3):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Tel Aviv
- South Korea (4):
  - Research Site, Cheongju-si
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Donostia / San Sebastian
  - Research Site, Granada
  - Research Site, Madrid
- Taiwan (2):
  - Research Site, Tainan
  - Research Site, Taipei
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Chiang Rai
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
- Turkey (Türkiye) (2):
  - Research Site, Ankara
  - Research Site, Yenimahalle
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual participant-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Aredo JV, Peled N, Arriola E, Wakelee H, Ahn MJ, Kwint MH, Taylor R, van der Gronde T, Nasirova F, Chen M. Osimertinib before and after chemoradiotherapy for unresectable stage III EGFR-mutated NSCLC: NEOLA Trial Protocol. Future Oncol. 2025 Dec;21(29):3731-3737. doi: 10.1080/14796694.2025.2587569. Epub 2025 Nov 14. PMID 41236484